CLINICAL TRIAL: NCT05850767
Title: The Effect of Sleep Deprivation on Passive Function, Active Function and Distance Modulation of the Vestibulo-Ocular Reflex
Brief Title: The Effect of Sleep Deprivation on Passive and Active Functions and Distance Modulation of the Vestibulo-Ocular Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yoav Gimon (Other)
Responsible Party: Sponsor-Investigator, Yoav Gimon, Senior lecturer, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 206/22
Record Dates: First submitted 2023-04-30; First posted 2023-05-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: VOR,vergence modulation,sleep deprivation,adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep deprivation (Experimental): Participants will stay fully awake for 24 hours.
  Interventions: Other: Sleep deprivation
- Normal sleep (No Intervention): Participant will sleep a normal night sleep.

INTERVENTIONS:
Other: Sleep deprivation — Participants will stay fully awake for 24 hours
  Arms: Sleep deprivation

SUMMARY:
The goal of this cross-over clinical trial is to evaluate the effect of 24 hours sleep deprivation on the Vestibulo-Ocular Reflex (VOR) in healthy participants.

The main questions it aims to answer are:

1. The effect of sleep deprivation on vestibular function.
2. The difference between passive and active VOR function following sleep deprivation.
3. The vergence mediated modulation ability of the VOR following sleep deprivation.
4. The effect of sleep deprivation on behavioral VOR function.

Participants will be tested before and after a normal night sleep and during 24 hours of sleep deprivation.

DETAILED DESCRIPTION:
The study will include two sleep protocols: Normal sleep and 24h sleep deprivation. The participants will be informed and will sign a consent form. Participants will then be randomly divided to begin with one of the sleep protocols. To avoid major changes in participants lifestyle, that might intervene with the basic measurements, both nights will take place within a maximum of one month and a minimum of one week for recovery between them. One week prior to each condition, participants will fill a sleep diary which will include their sleep duration to ensure that a routine sleep pattern will be maintained prior to each of the tests. Participants will be instructed not to consume alcoholic drinks or mind-altering substances for 24h prior, and during both conditions, and caffeine for 12h prior and during both conditions.

To enable normal sleep as possible, the normal sleep protocol will take place in each of the participants home. Matching environmental conditions will be kept to those of the clinic (lighting, white background) where the sleep deprivation protocol will be held. The participants will be tested using the Video Head Impulse test (vHIT) and the Computerized Dynamic Visual Acuity test (c-DVA) during both nights. The participants will be equipped with an ActiGraph watch wGT3X-BT to assure sleeping conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years old
* Healthy
* Persons who are not night shift workers
* Persons who are not used to but can keep awake for 24 hours

Exclusion Criteria:

* Night shift workers
* Vestibular system deficiency in vHIT test
* Active neurological disease
* Any orthopedic deficit in the cervical area preventing a proper vHIT examination
* A diagnosed sleep disorder or >5 score in the Pittsburgh sleep quality questionnaire Hebrew version (PSQI)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
VOR gain | 9pm before and 6am after normal sleep. 9pm, 2am and 6am during sleep deprivation.
  The calculated ratio between eye velocity and head velocity during brief head movements

SECONDARY OUTCOMES:
Logarithm of the Minimum Angle of Resolution (logMAR) | 6am following normal sleep and 6am during sleep deprivation.
  Units measuring visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Gimmon, Phd, Principal Investigator — University of Haifa, Haifa, Israel
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Chang TP, Schubert MC. Convergence Vestibulo-ocular Reflex in Unilateral Vestibular Hypofunction: Behavioral Evidence in Support of a Novel Gaze Stability Exercise. J Neurol Phys Ther. 2021 Jan;45(1):3-11. doi: 10.1097/NPT.0000000000000335. PMID 33065632